CLINICAL TRIAL: NCT00569959
Title: Assessment of Non-Fasting vs. Fasting Lipid Measures in Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 03363-05-A
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes Mellitus; Normal Glucose Metabolism; Hyperlipidemia
Keywords: fasting lipid measures; non-fasting lipid measures; clinical decision-making; LDL-Cholesterol
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting (Other)
  Interventions: Other: fasting 12+ hours
- Non-fasting (Other)
  Interventions: Other: Non-fasting

INTERVENTIONS:
Other: fasting 12+ hours — fasting 12+ hours
  Arms: Fasting
Other: Non-fasting — Non-fasting
  Arms: Non-fasting

SUMMARY:
This study will examine whether fasting and non-fasting lipid measures can provide similar clinical information in order to guide lipid management by primary physicians. It will compare fasting vs. non-fasting lipid measurements in patients with and without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Park Nicollet Health Services patients due for routine lipid measures

Exclusion Criteria:

* Unwilling or unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
LDL-Cholesterol | Fasting 12+ hours vs. Non-fasting

SECONDARY OUTCOMES:
Other lipid parameters | Fasting 12+ hours vs. non-fasting

CONTACTS AND LOCATIONS:
Overall Officials: William Richards, MD, Principal Investigator — Park Nicollet Health Services
Locations (1):
- Park Nicollet Internal and Family Medicine Clinics, Minneapolis, Minnesota, United States